CLINICAL TRIAL: NCT01958450
Title: Comparitive Study of Efficacy and Safety Between Fractional Er:YAG Laser and Bipolar Radiofrequency Treatment for Acne Scar
Brief Title: Comparison of the Efficacy of Fractional Er:YAG Laser for Acne Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-1061
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Scar
Keywords: acne scar; Laser therapy; wound healing
MeSH Terms: conditions — Cicatrix | interventions — Lasers, Solid-State; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Er:YAG laser (Experimental): acne scar treatment using Er:YAG laser
  Interventions: Procedure: Er:YAG laser
- Bipolar radiofrequency with diode laser (Active Comparator): Bipolar radiofrequency with diode laser
  Interventions: Procedure: Bipolar radiofrequency with diode laser

INTERVENTIONS:
Procedure: Er:YAG laser — acne scar treatment using Er:YAG laser
  Arms: Er:YAG laser
Procedure: Bipolar radiofrequency with diode laser — acne scar treatment with bipolar radiofrequency combined with diode laser
  Arms: Bipolar radiofrequency with diode laser

SUMMARY:
Compare the efficacy of frational Er:YAG laser and that of bipolar frequency with diode laser treatment.

DETAILED DESCRIPTION:
In acne scar treatment, ablational laser would be superior to nonablative laser treatment. Frational Er:YAG laser treatment is a effective treatment plan for acne scar without severe adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* moderate acne scar

Exclusion Criteria:

* taking steroids, nonsteroidal antiinflammatory drug, and isotretinoin
* anyone who received acne scar procedures within 6 months
* underlying diabetes mellitus, keloid, or malignancy

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Global asessment of acne scar | 12 weeks
  5 point grading of acne scar

SECONDARY OUTCOMES:
ECCA | 12 weeks
  quantative assessement of acne scar
adverse effect assessment | 12 weeks
  adverse effect assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Suh, PhD, Study Chair — Department of Dermatology, Seoul National University College of Medicine; Seonguk Min, Msc, Principal Investigator — Department of Dermatology, Seoul National University College of Medicine
Locations (1):
- Department of Dermatology, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Kutlubay Z, Gokdemir G. Treatment of atrophic facial acne scars with the Er:YAG laser: a Turkish experience. J Cosmet Laser Ther. 2010 Apr;12(2):65-72. doi: 10.3109/14764171003706141. PMID 20331342